CLINICAL TRIAL: NCT07277517
Title: The Effect of Integrating Pain Neuroscience Education(PNE) With Conventional Physiotherapy on Pain and Functional Disability in Patients With Acute Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1404.530
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Acute Low-back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Conventional Physiotherapy Plus Pain Neuroscience Education (PNE)" (Experimental)
  Interventions: Other: routine physiotherapy + traditional patient education; Behavioral: pain neuroscience education
- "Conventional Physiotherapy With Routine Back-Care Education" (Active Comparator)
  Interventions: Other: routine physiotherapy + traditional patient education

INTERVENTIONS:
Other: routine physiotherapy + traditional patient education — Conventional Physiotherapy (Control Group)
  Participants in the control group will receive a baseline physiotherapy protocol, administered twice weekly for four weeks (8 sessions total). Each session includes:
  Soft Tissue Mobilization (40 minutes): Four specific myofascial release techniques targeting the low back and pelvic muscles (e.g., transverse sliding of lumbar muscles, thoracolumbar fascia release, quadratus lumborum release, iliopsoas release).
  Transcutaneous Electrical Nerve Stimulation (TENS) (30 minutes): Applied crosswise over the low back with parameters set at 100 Hz frequency and 300 µs pulse width, adjusted to a strong but comfortable sensory level.
  Additionally, this group receives two individual 50-minute sessions of standard physical hygiene and routine back care education to control for the time and attention given to the experimental group's Pain Neuroscience Education.
Behavioral: pain neuroscience education — The experimental group receives the same conventional physiotherapy as the control group, with the addition of PNE. This consists of two individual, face-to-face educational sessions (40-50 minutes each), delivered before the first and after the last physiotherapy session. The curriculum is based on established resources ("Explain Pain" and "Pain Neuroscience Education: Teaching People About Pain") and uses metaphors, examples, and slides to reconceptualize pain by explaining neurobiology, central sensitization, and the distinction between pain and tissue injury. Understanding is assessed using the revised Neurophysiology of Pain Questionnaire (rNPQ), and participants receive a booklet for reinforced learning at home.
  Arms: "Conventional Physiotherapy Plus Pain Neuroscience Education (PNE)"

SUMMARY:
Acute low back pain is one of the most common health problems in the world. Most people experience it at least once in their lives, and although many cases improve within a few weeks, a significant number of patients continue to struggle with pain, fear of movement, stress, and reduced daily function. These psychological factors-such as catastrophizing ("my back is damaged"), fear of movement ("if I move, it gets worse"), and avoidance behaviors-can slow recovery and increase the risk of the pain becoming chronic.

Pain Neuroscience Education (PNE) is a modern educational approach that teaches patients how pain actually works in the nervous system. Instead of focusing only on muscles and bones, PNE helps people understand how the brain interprets pain, why pain can persist even without serious injury, and how thoughts, emotions, and behaviors can influence the experience of pain. Research shows that PNE can reduce fear, improve movement, and help people participate better in rehabilitation-especially in chronic pain. However, there is very limited high-quality evidence about its effects in acute low back pain.

The purpose of this study is to determine whether adding Pain Neuroscience Education to routine physiotherapy can improve recovery in people with acute low back pain.

To do this, the investigators will conduct a single-blind randomized clinical trial with two groups of patients:

Control group: Receives conventional physiotherapy, including soft-tissue mobilization and TENS, along with routine patient education about posture and back care.

Intervention group: Receives the same physiotherapy plus two structured sessions of Pain Neuroscience Education, delivered individually using simple explanations, metaphors, and visual materials.

Both groups will receive eight treatment sessions over four weeks.

The investigators will measure several important outcomes before starting treatment and immediately after the 8th session, including:

Pain intensity

Functional disability

Pain catastrophizing

Fear-avoidance beliefs

Fear of movement (kinesiophobia)

The investigators' hypothesis is that patients who receive PNE in addition to routine physiotherapy will show greater reductions in pain, disability, fear, and catastrophizing compared to those receiving physiotherapy alone.

If proven effective, this approach could provide a simple, low-cost, and safe addition to physiotherapy that not only reduces pain but also prevents acute low back pain from turning into a chronic condition. This could help improve patients' quality of life and reduce the economic and healthcare burden caused by low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* A primary complaint of acute low back pain (defined as pain between the bottom of the ribs and the gluteal fold), with or without leg pain.
* Pain duration of less than 6 weeks.
* Absence of any "red flags" for serious spinal pathology (e.g., tumor, infection, fracture, cauda equina syndrome), as confirmed by an orthopedist or neurologist.

Exclusion Criteria:

* Low back pain lasting more than 3 months (chronic low back pain).
* History of spinal surgery within the past 3 years.
* Inability to read or understand Persian.
* Diagnosed cognitive impairments.
* Unwillingness to continue the treatment or study protocol.
* Diagnosed rheumatic, neurological, cardiac, metabolic, or respiratory diseases.
* Diagnosis of fibromyalgia, chronic fatigue syndrome, loss of skin sensation, or skin inflammation/swelling in the low back area.
* Presence or emergence of any "red flag" condition.
* Missing more than 3 consecutive treatment sessions.
* Previous participation in Pain Neuroscience Education sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | first session (day 1), end of 8th session (4 weeks)
  pain intensity which will be measured by Visual Analog Scale The scale is from 0 to 10. The closer the number is to 10, the more severe the pain is.
Oswestwry Disability Index | first session (day 1), end of 8th session (4 weeks)
  functional disability which will be measured by Oswestry Disability Index The scale is from 0 to 100 percentage. The closer the number is to 100, the more severe is the disability level.

SECONDARY OUTCOMES:
Tampa Scale Of Kinesiophobia | first session (day 1), end of 8th session (4 weeks)
  Kinesiophobia which will be measured by Tampa Scale Of Kinesiophobia The scale scores are between 17 to 68 and the score of 38 and more, shows high fear of movement.
Fear Avoidance Beliefs Questionnaire | first session (day 1), end of 8th session (4 weeks)
  Fear Avoidance Beliefs Which will be measured by Fear Avoidance Beliefs Questionnaire
Pain Catastrophizing Scale | first session (day 1), end of 8th session (4 weeks)
  Pain Catastrophizing which will be measured by Pain Catastrophizing Scale

CONTACTS AND LOCATIONS:
Locations (1):
- rehabilitation facility, Iran university of medical science, Tehran, Iran